CLINICAL TRIAL: NCT05333341
Title: Pain Care at Home to Amplify Function (Pain CHAMP)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000031092; 1RM1DA055310-01 (NIH)
Record Dates: First submitted 2022-04-11; First posted 2022-04-19 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use Disorder; Opioid Misuse; Chronic Pain
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCM (Active Comparator): TCM uses clinical pharmacists leading LTOT reassessment and, when indicated for underlying OUD, buprenorphine (BUP) initiation in consultation with a BUP-prescribing physician. Clinical pharmacists will lead LTOT reassessment and, when indicated for underlying OUD, buprenorphine (BUP) initiation in consultation with a BUP-prescribing physician.
  Interventions: Behavioral: TCM
- TCM plus COPES (Experimental): Participants in this arm will use TCM plus COPES that will augment the effectiveness of TCM alone.
  Interventions: Behavioral: TCM plus COPES

INTERVENTIONS:
Behavioral: TCM — TCM care is remotely-delivered and medium-term (up to 12 months), with the objective of improving CP and OUD/misuse symptoms primarily through medication management.
  Arms: TCM
Behavioral: TCM plus COPES — The COPES program will augment the effectiveness of TCM alone. COPES is a 12-week, Interactive Voice Response (IVR)-facilitated program of CBT for CP and common sequelae (depressive symptoms, sleep difficulties, low physical activity). Ongoing COPES engagement will be tracked by the COPES system. The primary components of the intervention are: 1) a self-help handbook containing the rationale and instructions for using ten pain self-management skills and their corresponding weekly skill practice goals; 2) a pedometer-facilitated walking program; 3) daily, automated IVR calls to collect pain interference, sleep quality, pedometer-measured step count, and adherence to the pain coping skill practice ratings; and 4) weekly, two to four minute pre-recorded, personalized therapist messages based on participant IVR-reported data.
  Arms: TCM plus COPES

SUMMARY:
This project aims to test simultaneously the effectiveness of telemedicine and collaborative management (TCM) vs. TCM plus Cooperative Pain Education and Self-Management (COPES) on patient level outcomes and the impact of site-tailored Implementation Facilitation to work toward long term opioid therapy dose reduction. Pain CHAMP is a patient-level randomized hybrid II effectiveness-implementation trial comparing TCM vs. TCM + COPES on the primary composite outcome of pain interference and OUD/misuse symptoms.

DETAILED DESCRIPTION:
Pain CHAMP is a patient-level randomized hybrid II effectiveness-implementation trial comparing TCM vs. TCM + COPES on the primary composite outcome of pain interference and OUD/misuse symptoms. The investigators have developed two evidence-based collaborative care interventions that use focused resources to assist primary care providers (PCPs) in meeting the two main challenges in managing care for patients on long-term opioid therapy (LTOT) with chronic pain (CP) and opioid use disorder (OUD)/misuse: 1) reassessment of LTOT and switch to medication for opioid use disorder (MOUD) as indicated and 2) ready access to evidence-based behavioral pain treatment. Both interventions are entirely virtual and thus serve the needs of many underserved populations. Telemedicine Collaborative Management (TCM) features clinical pharmacists leading LTOT reassessment and buprenorphine (BUP) initiation in consultation with a BUP-prescribing physician. The TCM model is effective in decreasing pain interference, achieving LTOT dose reduction, BUP initiation and continuation, and shows greater patient engagement than the more resource intensive Integrated Pain Team comparator arm. Cooperative Pain Education and Self-Management (COPES), a cognitive-behavioral therapy (CBT) program delivered via telehealth that improves pain interference, improves access to evidence-based behavioral pain treatment.

While TCM and COPES are established interventions, the additional value of COPES-as a behavioral CP intervention paired with the pharmacologic-focused TCM for chronic pain and LTOT misuse/OUD--has not been tested. To advance systems-level approaches to addressing co-occurring CP, LTOT and OUD/misuse, this study will make two important steps forward. First, the investigators will use a pragmatic approach and randomize at the site-level so all eligible patients will receive standard-of-care treatment. Second, the study will train PCPs in how to re-assume care of patients' post-collaborative care to maintain gains made during the intervention/s. To meet these goals, the team of investigators with expertise conducting high-impact CP and OUD research propose Pain Care at Home to Amplify Function (Pain CHAMP) a hybrid II trial to test simultaneously the effectiveness of TCM vs. TCM plus COPES on patient level outcomes and the impact of site-tailored Implementation Facilitation on successful uptake of each intervention with the following specific aims:

Aim 1: Compare the effectiveness of pharmacist-led TCM vs TCM plus COPES on the primary composite outcome of improved pain interference and opioid safety as measured by opioid misuse or opioid use disorder. As secondary outcomes, we will compare groups on alcohol use, anxiety, depression, and sleep.

Aim 2: Evaluate the effectiveness of Implementation Facilitation for TCM and COPES on Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) guided outcomes using mixed qualitative-quantitative methods.

Aim 3: Examine the cost-effectiveness of TCM plus COPES, relative to TCM, on the primary composite outcome.

This study receives support from and included in the HEAL Initiative (https://heal.nih.gov/).

ELIGIBILITY:
Inclusion Criteria:

Participants:

* Engaged in TCM intervention (with or without COPES)

Providers:

* Engaged with a participating study site

Exclusion Criteria:

Participants:

* Not engaged in TCM intervention

Providers:

* Not engaged with a participating study site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving improvement in pain interference with no evidence of OUD or misuse | 10 months
  Proportion of participants achieving both improvement in pain interference by using ≥ 1 point improvement in pain interference as measured by the PEG-3 scale and no evidence of OUD or misuse (score 0 on TAPS-2 opioid items and medical chart review shows no evidence).

SECONDARY OUTCOMES:
Mean change in anxiety using the Generalized Anxiety Disorder-2 (GAD-2) questionnaire | 10 months
  Mean change in anxiety post intervention using GAD-2 will be assessed at Day 0 and 6 months post-intervention (10 months). Generalized Anxiety Disorder-2 questionnaire is a 2-item validated questionnaire used to screen for anxiety with a range of scores from 0-3. A score of 3 is considered positive for anxiety with lower scores indicating no or mild anxiety.
Mean change in depression assessed using Patient Health Questionnaire-2 (PHQ-2) | 10 months
  Mean change in depression post intervention using PHQ-2 will be assessed at Day 0 and 6 months post-intervention (10 months). The PHQ-2 consists of the first two questions of the Patient Health Questionnaire-9 and asks about the frequency of depressed mood and anhedonia over the past two weeks. Each question is answered on a scale of 0-3 as follows: 0 = Not at all, 1 = Several days, 2 = More than half the days, 3 = Nearly every day. Score ranges from 0-6, with a score of 0-2 being negative for potential major depressive disorder and a score of 3 or more being positive for potential major depressive disorder.
Proportion of participants with high-risk alcohol use assessed using Alcohol Use Disorders Identification Test-C (AUDIT-C) | 10 months
  Proportion of participants with high-risk alcohol use using AUDIT-C will be assessed at 6 months post-intervention (10 months). The AUDIT-C consists of 3 questions posed to participants about consumption habits that quantifies alcohol misuse. Each question is answered on a scale of 0-4 and total scores range from 0-8. Total scores of 5 or more indicates high-risk alcohol use.
Mean change in sleep assessed using Brief Pain Inventory (BPI) sleep item | 10 months
  Mean change in sleep post intervention using BPI sleep item will be assessed at Day 0 and 6 months post-intervention (10 months). The BPI rapidly assesses the severity of pain and its impact on functioning. BPI asks the participant to rate how pain interferes with daily activities. The sleep item to be used asks, "Circle the one number that describes how, during the past week, pain has interfered with your sleep", with a scale of 1 to 10, where "0" indicates "does not interfere and "10" indicates "completely interferes".

OTHER OUTCOMES:
Proportion of participants that initiate COPES | End of TCM implementation (approximately 30 months after start)
  Proportion of participants initiating COPES among patients randomized to COPES. Ongoing COPES engagement will be tracked by the COPES system.
Proportion of participants on a TCM panel that achieve BUP stabilization | 12 months
  Proportion of eligible participants on a TCM panel achieving BUP stabilization defined as using BUP at least 70 of the final 90 days of the 12-month period following TCM intake assessed by the electronic pharmacy record review.
Proportion of PCP at each site that prescribed buprenorphine during the study period | End of TCM implementation (approximately 30 months after start)
  Proportion of PCP at each site that prescribed buprenorphine during the study period assessed by the electronic pharmacy record review.
Proportion of patient encounters in which individual TCM components were implemented over the intervention period | End of TCM implementation (approximately 30 months after start)
  Proportion of patient encounters in which individual TCM components were implemented by providers over the intervention using the participants electronic health record period to assess implementation.
Maintenance of medication management for ≥1 patients post-implementation | 6 months post TCM implementation
  Proportion of sites in which the TCM team maintained medication management for ≥1 patients post-implementation using the electronic pharmacy record.

CONTACTS AND LOCATIONS:
Overall Officials: William Becker, MD, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Little Rock VAMC, Little Rock, Arkansas
  - Eastern Colorado HCS, Aurora, Colorado
  - VA Connecticut HCS, West Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
A fully de-identified data set will be shared. The data shall exclude the following direct identifiers of the individual:
  (i) Names; (ii) Postal address information, other than town or city, State, and zip code; (iii) Telephone numbers; (iv) Fax numbers; (v) Electronic mail addresses; (vi) Social security numbers; (vii) Medical record numbers; (viii) Health plan beneficiary numbers; (ix) Account numbers; (x) Certificate/license numbers; (xi) Vehicle identifiers and serial numbers, including license plate numbers; (xii) Device identifiers and serial numbers; (xiii) Web Universal Resource Locators (URLs); (xiv) Internet Protocol (IP) address numbers; (xv) Biometric identifiers, including finger and voice prints; and (xvi) Full face photographic images and any comparable images. Additionally all dates of service and assessment will be masked.